CLINICAL TRIAL: NCT03594877
Title: Effectiveness of the Sublimated Mare Milk on the Gut Microbiome in Psoriasis and Healthy Patients
Brief Title: Effect of Sublimated Mare Milk Supplement on Gut Microbiome in Psoriasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: Eurasia Invest Ltd. (Industry); Ministry of Education and Science, Republic of Kazakhstan (Other Government); Centre for Dermatology and Sexually Transmitted Diseases, Astana, Kazakhstan (Unknown)
Responsible Party: Principal Investigator, Bakytgul Yermekbayeva, MD, PhD, Nazarbayev University Medical Center
Organization: Nazarbayev University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PsS.2017.1.1
Record Dates: First submitted 2018-06-25; First posted 2018-07-20 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Psoriasis
Keywords: mare milk; gut microbiome; psoriasis; immune markers
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psoriasis patients (Experimental): Patients with verified diagnosis of psoriasis would be given standard treatment for the first 3 months, and then followed with the standard therapy accompanied with the sublimated mare milk supplement for additional 3 months.
  Interventions: Dietary Supplement: Sublimated mare milk
- Healthy volunteers (No Intervention): Healthy patients will be enrolled in this study, and their gut microbiota composition as well as immune system indicators will be used for comparison with the psoriasis group.

INTERVENTIONS:
Dietary Supplement: Sublimated mare milk — The dietary supplement mare milk product, which is obtained from fresh (few hours) through sublimation process. This product is first mixed with warm water (37-38 degrees of Celsius) and then will be given to participants.
  Arms: Psoriasis patients

SUMMARY:
This study evaluates the effect of dietary supplement consisting of sublimated mare milk on intestinal microbiota among psoriasis and healthy participants.

DETAILED DESCRIPTION:
The gut microbiome is believed to play an important role in the immune system regulation, since intestines are the largest lymphoid organ in a human body. Deviations from healthy composition of intestinal flora are associated with various diseases including allergy and autoimmunity. Psoriasis is the one of the long-lasting autoimmune diseases that is characterized by patches on the skin and further health complications throughout the life. However, lack of studies does not allow proper evaluation of role of gut microbiome in psoriasis patients. Therefore, potential interplay between gut microbiome and immune system in psoriasis would be studied in this clinical trial. Particularly, the investigators hypothesize that sublimated mare milk supplement can have an impact on gut immune system and gut microbiome composition in the psoriasis patients.

In this trial, there will be two parallel groups: crossover psoriasis patients (standard treatment first for 3 months, next 3 months standard treatment plus sublimated mare milk supplement) and healthy volunteers group. Subsequently, association of intestinal flora with immune status will be analyzed and compared between these groups.

ELIGIBILITY:
Inclusion Criteria.

Inclusion criteria for experimental group:

* Patients with a verified diagnosis of moderate to severe psoriasis
* Aged 30 to 45 years
* Absence of an allergic reaction to dairy products
* Lack of prescription of antibacterial drugs for the last 3 months prior to admission
* Willingness to consent to participate in the study

Inclusion criteria for healthy volunteers group.

* Patients with no diagnosis of psoriasis
* Aged 30 to 45 years

Exclusion Criteria:

* Presence of chronic dermatoses, diseases of the organs of the gastrointestinal tract
* Presence of severe concomitant diseases of the kidneys, liver, cardiovascular, respiratory and other body systems, oncological, mental health and decompensated endocrine diseases, tuberculosis, and HIV infection
* Pregnancy and/or lactation
* Patient involvement in other clinical trials within the last 3 months
* Refusal to participate in the study

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in composition of microorganisms in stool after the supplement intervention. | Baseline, 6 weeks, 12 weeks
  Change in composition of intestinal microbiota will be determined comparing with the baseline results using DNA sequencing Illumina MiSeq System.
Change from baseline of biomarkers of inflammation in intestines. | Baseline, 6 weeks, 12 weeks
  The change of immunity will be evaluated from stool specimens according to baseline results of inflammatory cytokines, interleukins, and antibodies. Number of patients, in whom change is statistically significant, will be reported in the results.

SECONDARY OUTCOMES:
PASI index for psoriasis | Baseline & 12 weeks
  Dermatological status of PASI index will be evaluated according to the international protocols for treatment of psoriasis (NICE guidance).
Change from baseline in Vitamin D levels | Baseline & 12 weeks
  Blood levels of Vitamin D will be compared between baseline and later periods in psoriasis patients.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center, Kazakhstan, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung I, Garrett JP, Shahane A, Kwan M. Do bugs control our fate? The influence of the microbiome on autoimmunity. Curr Allergy Asthma Rep. 2012 Dec;12(6):511-9. doi: 10.1007/s11882-012-0291-2. PMID 22886439
- [Background] Ely PH. Is psoriasis a bowel disease? Successful treatment with bile acids and bioflavonoids suggests it is. Clin Dermatol. 2018 May-Jun;36(3):376-389. doi: 10.1016/j.clindermatol.2018.03.011. Epub 2018 Mar 28. PMID 29908580
- [Background] Yan D, Issa N, Afifi L, Jeon C, Chang HW, Liao W. The Role of the Skin and Gut Microbiome in Psoriatic Disease. Curr Dermatol Rep. 2017 Jun;6(2):94-103. doi: 10.1007/s13671-017-0178-5. Epub 2017 Apr 22. PMID 28804689
- [Background] Scher JU, Ubeda C, Artacho A, Attur M, Isaac S, Reddy SM, Marmon S, Neimann A, Brusca S, Patel T, Manasson J, Pamer EG, Littman DR, Abramson SB. Decreased bacterial diversity characterizes the altered gut microbiota in patients with psoriatic arthritis, resembling dysbiosis in inflammatory bowel disease. Arthritis Rheumatol. 2015 Jan;67(1):128-39. doi: 10.1002/art.38892. PMID 25319745
- [Background] Gao Z, Tseng CH, Strober BE, Pei Z, Blaser MJ. Substantial alterations of the cutaneous bacterial biota in psoriatic lesions. PLoS One. 2008 Jul 23;3(7):e2719. doi: 10.1371/journal.pone.0002719. PMID 18648509
- [Background] Codoner FM, Ramirez-Bosca A, Climent E, Carrion-Gutierrez M, Guerrero M, Perez-Orquin JM, Horga de la Parte J, Genoves S, Ramon D, Navarro-Lopez V, Chenoll E. Gut microbial composition in patients with psoriasis. Sci Rep. 2018 Feb 28;8(1):3812. doi: 10.1038/s41598-018-22125-y. PMID 29491401
- [Background] Eppinga H, Sperna Weiland CJ, Thio HB, van der Woude CJ, Nijsten TE, Peppelenbosch MP, Konstantinov SR. Similar Depletion of Protective Faecalibacterium prausnitzii in Psoriasis and Inflammatory Bowel Disease, but not in Hidradenitis Suppurativa. J Crohns Colitis. 2016 Sep;10(9):1067-75. doi: 10.1093/ecco-jcc/jjw070. Epub 2016 Mar 12. PMID 26971052
- [Result] Yegorov S, Babenko D, Kozhakhmetov S, Akhmaltdinova L, Kadyrova I, Nurgozhina A, Nurgaziyev M, Good SV, Hortelano GH, Yermekbayeva B, Kushugulova A. Psoriasis Is Associated With Elevated Gut IL-1alpha and Intestinal Microbiome Alterations. Front Immunol. 2020 Oct 1;11:571319. doi: 10.3389/fimmu.2020.571319. eCollection 2020. PMID 33117362
- [Result] Togzhan Algazina, Alexandr Gulyayev, Alma Aimoldina, Almagul Kushugulova, Bakytgul Yermekbayeva*. Clinical assessment of the use of sublimated mare's milk in complex therapy of mild and moderate psoriasis // Journal of Global Pharma Technology.- 2020.- Vol.12.- Issue 06.- P. 18-25